CLINICAL TRIAL: NCT04404998
Title: Lunch Meal Study for Men and Women
Brief Title: The Influence of Energy Density and Information on Meal Intake in Adults
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Issues with recruitment due to COVID 19
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Barbara J. Rolls, Professor of Nutrition and Director of the Laboratory for the Study of Human Ingestive Behavior, Penn State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: FoodED601
Record Dates: First submitted 2020-03-11; First posted 2020-05-28 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Feeding Behavior
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Lower Energy Density & Lower Satiation (Experimental): Test meal with lower energy density and lower satiation information
  Interventions: Other: Lower Energy Density; Other: Lower Satiation
- Lower Energy Density & Higher Satiation (Experimental): Test meal with lower energy density and higher satiation information
  Interventions: Other: Lower Energy Density; Other: Higher Satiation
- Higher Energy Density & Lower Satiation (Experimental): Test meal with higher energy density and lower satiation information
  Interventions: Other: Higher Energy Density; Other: Lower Satiation
- Higher Energy Density & Higher Satiation (Experimental): Test meal with higher energy density and higher satiation information
  Interventions: Other: Higher Energy Density; Other: Higher Satiation

INTERVENTIONS:
Other: Lower Energy Density — Test meal with lower energy density
  Arms: Lower Energy Density & Higher Satiation; Lower Energy Density & Lower Satiation
Other: Higher Energy Density — Test meal with higher energy density
  Arms: Higher Energy Density & Higher Satiation; Higher Energy Density & Lower Satiation
Other: Lower Satiation — Information on lower satiation
  Arms: Higher Energy Density & Lower Satiation; Lower Energy Density & Lower Satiation
Other: Higher Satiation — Information on higher satiation
  Arms: Higher Energy Density & Higher Satiation; Lower Energy Density & Higher Satiation

SUMMARY:
The purpose of this study is to gain a better understanding of how energy density and cognitive framing of satiation using food information can influence consumption at a meal. This study also aims to investigate the influence of energy density and food information on sensory specific satiety (the decline in the subjective pleasantness of a food as it is eaten).

ELIGIBILITY:
Inclusion Criteria:

* Ability to attend all test meals
* Be fully vaccinated against COVID-19
* Regularly eat 3 meals/day
* Being willing to avoid alcohol the day before and during test days
* Have a body mass index greater than 18.0 kg/meters squared
* Being willing to refrain from eating after 10 pm the evening before test sessions

Exclusion Criteria:

* Being a smoker
* Being an athlete in training
* Being pregnant or breastfeeding at the time of screening
* Have taken prescription or non-prescription drugs that may affect appetite or food intake within the last 3 months
* Dislike or inability to eat the test foods
* Currently dieting to gain or lose weight
* Have a health condition that affects appetite
* Have participated in a similar study in our lab in the past year
* Being a student, faculty, or staff member in nutritional sciences or psychology

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2021-08-03 (Actual); Primary Completion 2021-11-08 (Actual); Study Completion 2021-11-08 (Actual)

PRIMARY OUTCOMES:
Change in food intake by weight | Weeks 1, 2, 3, 4
  Weight of food consumed measured in grams (g)
Change in energy intake | Weeks 1, 2, 3, 4
  Energy content of food consumed measured in kilocalories (kcal)

SECONDARY OUTCOMES:
Change in palatability rating of food samples | Weeks 1, 2, 3, 4
  Difference between post-meal and pre-meal palatability of the food samples measured by Visual Analogue Scales (ranging from 0 mm to 100 mm) to assess Sensory-Specific Satiety
Change in prospective consumption rating of food samples | Weeks 1, 2, 3, 4
  Difference between post-meal and pre-meal prospective consumption of food samples measured by Visual Analogue Scales (ranging from 0 mm to 100 mm) to assess Sensory-Specific Satiety
Change in hunger rating | Weeks 1, 2, 3, 4
  Difference between post-meal and pre-meal hunger measured by Visual Analogue Scales (ranging from 0 mm to 100 mm)
Change in fullness rating | Weeks 1, 2, 3, 4
  Difference between post-meal and pre-meal fullness measured by Visual Analogue Scales (ranging from 0 mm to 100 mm)
Change in test meal prospective consumption rating | Weeks 1, 2, 3, 4
  Difference in prospective consumption measured by Visual Analogue Scales (ranging from 0 mm to 100 mm)
Change in test meal fillingness rating | Weeks 1, 2, 3, 4
  Difference in fillingness measured by Visual Analogue Scales (ranging from 0 mm to 100 mm)
Change in test meal palatability rating | Weeks 1, 2, 3, 4
  Difference in palatability of the test meal measured by Visual Analogue Scales (ranging from 0 mm to 100 mm)
Change in estimation of proportion of test meal consumed | Weeks 1, 2, 3, 4
  Difference in estimation of proportion of test meal consumed measured by Visual Analogue Scales (ranging from 0 mm to 100 mm)
Change in estimation of energy content of test meal consumed | Weeks 1, 2, 3, 4
  Difference in estimation of energy content of test meal consumed measured by Visual Analogue Scales (ranging from 0 mm to 100 mm)

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratory for the Study of Human Ingestive Behavior, The Pennsylvania State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No